CLINICAL TRIAL: NCT05555602
Title: Clinical Observation of the Comfort and Efficacy of Carbon Dioxide(CO2) Laser 10,600 nm Combined With Cold-air Cooling Device Zimmer Cryo 6 for Burn Scars or Linear Scars.
Brief Title: Observation of the Comfort and Efficacy of CO2 Laser Combined With Cryo 6 for Burn or Linear Scars.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaiyang Lv, MD-PhD (Other)
Collaborators: Zimmer Medical Devices (Shanghai) Co., Ltd. (Unknown)
Responsible Party: Sponsor-Investigator, Kaiyang Lv, MD-PhD, Associate Chief Physician, Associate Professor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: XH-21-010
Record Dates: First submitted 2021-11-16; First posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Cryotherapy Effect; Burn Scar; Scar; Previous Cesarean Section
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control group: CO2 fractional laser alone (No Intervention): This group of patients is the treatment control group. During the treatment period, the cold-air cooling device Cryo 6 will be placed next to the laser equipment but not started. The air outlet position is about 3 to 7 centimeters away from the skin, and it will move slowly and synchronously according to the laser position. The skin temperature will be synchronously monitored and recorded by hand-held infrared thermometry. After the operation, the investigators use hospital's routine aftercare procedures, and continue to use hand-held infrared thermometry to synchronously monitor the skin temperature.
- Combination group: CO2 fractional laser combined with Cryo 6 (Experimental): During the CO2 fractional laser treatment, cool the skin with cold-air cooling device Cryo 6. Set the wind to level 5, and the maximum time to 30 minutes. The air outlet position is about 3 to 7 centimeters away from the skin, and it will move slowly and synchronously according to the laser position. The skin temperature will be synchronously monitored by hand-held infrared thermometry and maintained at 0°C to 5°C. After the operation, the investigators use hospital's routine aftercare procedures and cooling with Cryo 6 on the skin synchronously. The wind level can be selected by patients themselves from level 3 to 7, and the time can be set for 5 minutes. Put the air outlet about 3 to 7 centimeters away from the skin, and move it slowly and dynamically in this area of skin to monitor and record the skin temperature synchronously.
  Interventions: Device: Cold-air cooling

INTERVENTIONS:
Device: Cold-air cooling — Cryo 6 works with a compressor system like those in refrigerators and uses ambient air to generate a permanent stream of cold air with a maximum flow to 1000 L/min and a temperature as low as -30°C, depending on the cooling delivery system and the desired cooling level (range 1-9).
  Other Names: Zimmer MedizinSysteme Cryo 6
  Arms: Combination group: CO2 fractional laser combined with Cryo 6

SUMMARY:
To investigate the effect of 10,600 nm CO2 laser combined with Zimmer Cryo 6 forced cold air device on the comfort and efficacy of patients with burn scars or post-operative linear scars, and to provide a safer, more effective and more satisfactory program for clinical treatment of burn scars or post-operative linear scars.

DETAILED DESCRIPTION:
Objective: To investigate the effect of 10,600 nm CO2 laser combined with the cold-air cooling device Zimmer Cryo 6 on the comfort and efficacy of patients with burn scars or post-operative linear scars, and to provide a safer, more effective and more satisfactory program for clinical treatment of burn scars or post-operative linear scars.

Secondary objective: To investigate the adverse effects of the cold-air cooling device Zimmer Cryo 6 in combination with the 10,600 nm CO2 fractional laser treatment for patients with burn scars or post-operative linear scars.

ELIGIBILITY:
Inclusion Criteria:

1. Age 14-60 years;
2. The patient agreed to participate in the experiment and signed the informed consent by himself/herself or his/her legal representative;
3. The clinical diagnosis was burn scar or post-operative linear scar, and the total area was more than 5 cm2.
4. No other treatment such as laser or chemical exfoliation was performed on the lesion within the recent half year.
5. Skin lesions were free of bleeding, ulceration, infection and other conditions affecting the visual field of laser treatment.

Exclusion Criteria:

1. Patients with an active or established sun tan;
2. Patients with history of allergic reaction to to topical anesthesia;
3. Patients with history of keloid scarring, abnormal wound healing and/or prone to bruising;
4. Skin malignant tumors or precancerous lesions;
5. Patients with diabetes, heart disease, epilepsy, connective tissue disease, etc.;
6. Pregnant or breastfeeding patients;
7. Patients with recent skin infections (such as viral and bacterial infections);
8. Patients who are using other methods to treat similar diseases;
9. Patients who had taken isotretinoin within the past year;
10. History of cryoglobulinaemia;
11. History of cold agglutinin disease and cold haemolysis;
12. History of cold urticaria;
13. Parts of the body with impaired circulation;
14. Raynaud's disease;
15. Parts of the body with impaired sensitivity;
16. Trophic disorders;
17. Hypersensitivity to cold;
18. Patients with mental illness;
19. Other ineligible patients.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-23 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) | Immediately after treatment
  The Numeric Rating Scale (NRS) is a numbered version of the Visual Analog Pain Scale (VAS) in which the patient can select one number that best describes the pain. Scale from minimum "0" to maximum "10" for total 11 integers. "0" represents no pain, and "10" represents worst pain imaginable.

SECONDARY OUTCOMES:
Skin temperature | Baseline, immediately after treatment
  The skin temperature will be monitored and recorded by hand-held infrared thermometry.
Number of treatment interruptions | Immediately after treatment
  The physician calculates the number of interruptions that the patient calls off during treatment.

OTHER OUTCOMES:
Scar area | Baseline, 1 month after the 1st treatment, 1 month after the 2nd treatment, 1 month after the 3rd treatment
  Analyze the scar pattern using Antera 3D software for Scar area (cm2).
Scar color | Baseline, 1 month after the 1st treatment, 1 month after the 2nd treatment, 1 month after the 3rd treatment
  Analyze the scar pattern using Antera 3D software for scar color (CIE L*a*B*).
Scar volume | Baseline, 1 month after the 1st treatment, 1 month after the 2nd treatment, 1 month after the 3rd treatment
  Analyze the scar pattern using Antera 3D software for scar volume (cm3).
Scar melamin | Baseline, 1 month after the 1st treatment, 1 month after the 2nd treatment, 1 month after the 3rd treatment
  Analyze the scar pattern using Antera 3D software for scar melanin.
Scar erythema | Baseline, 1 month after the 1st treatment, 1 month after the 2nd treatment, 1 month after the 3rd treatment
  Analyze the scar pattern using Antera 3D software for scar erythema.
Satisfaction evaluation | 1 month after the 1st and the 3rd treatments.
  The patients were rated as very dissatisfied, dissatisfied, fair, satisfied, and very satisfied with the improvement of scars.

CONTACTS AND LOCATIONS:
Overall Officials: Yo-Yu Tseng, M.Sc, Principal Investigator — Zimmer Medical Devices (Shanghai) Co., Ltd.
Locations (1):
- Xinhua Hospital affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tian H, Wang L, Xie W, Shen C, Guo G, Liu J, Han C, Ren L, Liang Y, Tang Y, Wang Y, Yin M, Zhang J, Huang Y. Epidemiologic and clinical characteristics of severe burn patients: results of a retrospective multicenter study in China, 2011-2015. Burns Trauma. 2018 May 23;6:14. doi: 10.1186/s41038-018-0118-z. eCollection 2018. PMID 29850643
- [Background] Waibel J, Beer K. Ablative fractional laser resurfacing for the treatment of a third-degree burn. J Drugs Dermatol. 2009 Mar;8(3):294-7. PMID 19271380
- [Background] Kwan JM, Wyatt M, Uebelhoer NS, Pyo J, Shumaker PR. Functional improvement after ablative fractional laser treatment of a scar contracture. PM R. 2011 Oct;3(10):986-7. doi: 10.1016/j.pmrj.2011.07.007. No abstract available. PMID 22024331
- [Background] Kineston D, Kwan JM, Uebelhoer NS, Shumaker PR. Use of a fractional ablative 10.6-mum carbon dioxide laser in the treatment of a morphea-related contracture. Arch Dermatol. 2011 Oct;147(10):1148-50. doi: 10.1001/archdermatol.2011.247. No abstract available. PMID 22006130
- [Background] Haedersdal M. Fractional ablative CO(2) laser resurfacing improves a thermal burn scar. J Eur Acad Dermatol Venereol. 2009 Nov;23(11):1340-1. doi: 10.1111/j.1468-3083.2009.03215.x. Epub 2009 Mar 4. No abstract available. PMID 19309424
- [Background] Bowen RE. A novel approach to ablative fractional treatment of mature thermal burn scars. J Drugs Dermatol. 2010 Apr;9(4):389-92. PMID 20514799
- [Background] Tierney EP, Hanke CW. The effect of cold-air anesthesia during fractionated carbon-dioxide laser treatment: Prospective study and review of the literature. J Am Acad Dermatol. 2012 Sep;67(3):436-45. doi: 10.1016/j.jaad.2011.01.026. Epub 2012 Jun 12. PMID 22695102
- [Background] Altshuler GB, Zenzie HH, Erofeev AV, Smirnov MZ, Anderson RR, Dierickx C. Contact cooling of the skin. Phys Med Biol. 1999 Apr;44(4):1003-23. doi: 10.1088/0031-9155/44/4/014. PMID 10232811
- [Background] Chess C, Chess Q. Cool laser optics treatment of large telangiectasia of the lower extremities. J Dermatol Surg Oncol. 1993 Jan;19(1):74-80. doi: 10.1111/j.1524-4725.1993.tb03331.x. PMID 8454790
- [Background] Gilchrest BA, Rosen S, Noe JM. Chilling port wine stains improves the response to argon laser therapy. Plast Reconstr Surg. 1982 Feb;69(2):278-83. doi: 10.1097/00006534-198202000-00017. PMID 7054797
- [Background] Kelly KM, Nelson JS, Lask GP, Geronemus RG, Bernstein LJ. Cryogen spray cooling in combination with nonablative laser treatment of facial rhytides. Arch Dermatol. 1999 Jun;135(6):691-4. doi: 10.1001/archderm.135.6.691. PMID 10376697
- [Background] Kim J, Shin W. How to do random allocation (randomization). Clin Orthop Surg. 2014 Mar;6(1):103-9. doi: 10.4055/cios.2014.6.1.103. Epub 2014 Feb 14. PMID 24605197
- [Background] Matias AR, Ferreira M, Costa P, Neto P. Skin colour, skin redness and melanin biometric measurements: comparison study between Antera((R)) 3D, Mexameter((R)) and Colorimeter((R)). Skin Res Technol. 2015 Aug;21(3):346-62. doi: 10.1111/srt.12199. Epub 2015 Feb 3. PMID 25645051
- [Background] Handford C, Buxton P, Russell K, Imray CE, McIntosh SE, Freer L, Cochran A, Imray CH. Frostbite: a practical approach to hospital management. Extrem Physiol Med. 2014 Apr 22;3:7. doi: 10.1186/2046-7648-3-7. eCollection 2014. PMID 24764516
- [Background] McIntosh SE, Opacic M, Freer L, Grissom CK, Auerbach PS, Rodway GW, Cochran A, Giesbrecht GG, McDevitt M, Imray CH, Johnson EL, Dow J, Hackett PH; Wilderness Medical Society. Wilderness Medical Society practice guidelines for the prevention and treatment of frostbite: 2014 update. Wilderness Environ Med. 2014 Dec;25(4 Suppl):S43-54. doi: 10.1016/j.wem.2014.09.001. PMID 25498262
- [Result] Raulin C, Grema H. Single-pass carbon dioxide laser skin resurfacing combined with cold-air cooling: efficacy and patient satisfaction of a prospective side-by-side study. Arch Dermatol. 2004 Nov;140(11):1333-6. doi: 10.1001/archderm.140.11.1333. PMID 15545541